CLINICAL TRIAL: NCT02284607
Title: A PHASE I, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, SINGLE-ASCENDING DOSE STUDY TO INVESTIGATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF HIGH DOSE MHAA4549A IN HEALTHY VOLUNTEERS
Brief Title: A Study of High Dose MHAA4549A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GV29609
Record Dates: First submitted 2014-10-31; First posted 2014-11-06 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gedivumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MHAA4549A higher dose (Experimental)
  Interventions: Drug: MHAA4549A
- MHAA4549A lower dose (Experimental)
  Interventions: Drug: MHAA4549A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHAA4549A — MHAA4549A single, intravenous dose administration, lower dose level
  Arms: MHAA4549A lower dose
Drug: MHAA4549A — MHAA4549A single, intravenous dose administration, higher dose level
  Arms: MHAA4549A higher dose
Drug: Placebo — Matching placebo to MHAA4549A administration
  Arms: Placebo

SUMMARY:
This Phase 1, randomized, double-blind, placebo-controlled study will evaluate the safety, tolerability and pharmacokinetics of two, single intravenous (IV) high doses of MHAA4549A as compared to placebo when administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive
* Weight 40 - 100 kg
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, vital signs, and clinical laboratory evaluations
* Willing to use acceptable contraceptive measures as defined by the protocol
* Agreeable to, and deemed able to by the investigator, to comply with the requirements of the study, including the follow-up period
* Willing to abstain from the use of drugs of abuse while enrolled in the study

Exclusion Criteria:

* History or clinically significant manifestations of disorders
* History of acute allergic reaction or drug allergies
* History or presence of an abnormal ECG
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit
* History of significant drug abuse within 1 year prior to screening
* Current tobacco smokers
* Positive drug screen at screening or at check-in
* Positive pregnancy test result at screening or Day -1 or breast feeding during the study
* Males who have a pregnant female partner
* Donation of plasma within 7 days prior to study drug administration
* Donation or loss of whole blood
* Receipt of blood products within 2 months before initiation of dosing on Day 1
* History of malignancy within 10 years of screening except completely excised basal cell carcinoma or squamous cell carcinoma of the skin
* History of severe systemic bacterial, fungal, or parasitic infections associated with more than two hospitalizations per year or more than two courses of intravenous (IV) antibiotics within 1 year
* Received oral antibiotics within 4 weeks before initiation of dosing on Day 1, or IV antibiotics within 8 weeks before initiation of dosing
* Hospitalization within 4 weeks before initiation of dosing on Day 1
* Use of any over the counter or prescription medications/products within 7 days prior to Day 1 and unwilling to abstain from the use of such drugs up until at least the Day 29 study visit, unless deemed acceptable by the investigator and Sponsor
* Participation in a clinical trial within 4 weeks
* Received any vaccine within 14 days prior to screening
* Positive blood test for chronic viral infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of adverse events (AEs) | Until study discontinuation/termination, up to 120 days
Changes in vital signs during and following MHAA4549A administration | From baseline to end of study, up to 120 days
Changes in ECG findings during and following MHAA4549A administration | From baseline to end of study, up to 120 days
Severity of AEs | Until study discontinuation/termination, up to 120 days

SECONDARY OUTCOMES:
Pharmacokinetics (composite outcome measure): parameters derived from the nasal and serum concentration-time profile of MHAA4549A (area under the concentration-time curve [AUC], Cmax, tmax, clearance, Vss, half-life (t1/2), mean residence time) | Up to 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- inVentiv Health Clinique, Québec, Quebec, Canada

REFERENCES:
- [Derived] Lim JJ, Deng R, Derby MA, Larouche R, Horn P, Anderson M, Maia M, Carrier S, Pelletier I, Burgess T, Kulkarni P, Newton E, Tavel JA. Two Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Studies To Investigate the Safety, Tolerability, and Pharmacokinetics of an Anti-Influenza A Virus Monoclonal Antibody, MHAA4549A, in Healthy Volunteers. Antimicrob Agents Chemother. 2016 Aug 22;60(9):5437-44. doi: 10.1128/AAC.00607-16. Print 2016 Sep. PMID 27381392